CLINICAL TRIAL: NCT03128450
Title: A Single Arm, Open-Label，Pilot Study to Evaluate the Safety and Efficacy of Human Neural Stem Cells Injection (ANGE-S003) Through Nasal Way Delivery to Patients With Parkinson's Disease
Brief Title: A Study To Evaluate the Safety and Efficacy of Human Neural Stem Cells for Parkinson's Disease Patient
Acronym: hNSCPD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Second Affiliated Hospital
Record Dates: First submitted 2017-02-09; First posted 2017-04-25 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Neural stem cell; Nasal delivery
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- h-NSC arm (Experimental): human neural stem cell: 100ul/vessel，2 vessel/one bag，≥2×10 6cells/vessel，produced by Shanghai Angecon Biotechology Cooperate.
  One enrolled PD patient was given 2 vessels h-NSC througth nasal cavity weekly for 4 weeks。Total cell number will be over ≥4×10 6cells for one time.
  Interventions: Biological: human neural stem cell

INTERVENTIONS:
Biological: human neural stem cell — human neural stem cell: 100ul/vessel，2 vessel/one bag，≥2×10 6cells/vessel

SUMMARY:
This Pilot study will evaluate the safety and Efficacy of an investigational cell transplantation therapy, h-NSC, in patients with Parkinson's disease, through nasal drug delivery, a new delivery way. All patients will receive the therapy, which consists of human neural stem cells,

DETAILED DESCRIPTION:
h-NSC is a cellular therapeutic consisting of human fetal neural stem cells (h-NSC). h-NSC injection will be delivered through nasal way for patients with Parkinson's disease (PD).

The study will enroll 12 moderate to severe PD patients to be treated with the cell injection therapy at the same dose. The total therapy course will be four weeks，one dose for one week. The follow up will be two times within 24 weeks after finishing the treatment. The main objective of the study is to evaluate the efficacy and safety of the cell transplantation by this new delivery way.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with idiopathic PD, at least with two key symptoms (Static tremor, bradykinesia, rigidity ) , without any other evidence of Secondary Parkinson's syndrome.
* Disease course ≥7 years，modified Hoehn-Yahr is 3-5 stage
* Patient age ≥35 years
* Patients receiving a stable dose of levodopa for at least 1 months with the expectation that the treatment will remain unchanged throughout the course of the study
* The doses of levodopa ≥300mg •Signed informed consent form (ICF) by patient self or his law-in relationship before enrollment.

Exclusion Criteria:

* Hepatic dysfunction(transaminase ≥1.5 normal range), Renal dysfunction(Cr>2.0mg/dl or 177μmol/L)，Cardiac dysfunction or other severe systematic diseases etc.
* Suffering malignancy or during anti-cancer treatment period.
* Pregancy, lactation or possible pregancy and plan to pregancy patient
* Attended other intervention clinical trial within 3 months aftre getting ICF, or during other ongoing intervention clinical trial
* Investigator think inappropriate patient for this protocol

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Unified Parkinson's Disease Reting Scale(UPDRS)score from baseline | Baseline and 16, 28 weeks
  Improvement rate of UPDRS motor score defined as below:
  Reduction rate =（baseline score 16, 28 weeks score after therapy）/ baseline score×100%.
  Based on reduction rate, the efficacy can be defined as complete remission, partial remission, effective and invalid The reduction rate will be 100%, >50%, >25-50%, ≤ 25% for complete remission, partial remission, effective and invalid.
  The improvement rate =[(complete+partial+effective patient number)/total patient number]×100％

SECONDARY OUTCOMES:
motor function index | baseline and 16, 28 weeks
  Hoehn-Yahr modified score
Non-motor function score:cognitive function | baseline and 16, 28 weeks
  Minimum Mental State Examination and Montreal Cognitive Assessment to assess cognitive function
Non-motor function score:smell | baseline and 16, 28 weeks
  Argentina Hyposmia Rating Scales is used to detect the smell
Non-motor function score:fatigue | baseline and 16, 28 weeks
  Fatigue Severity Scale to assess the extent of fatigue
Non-motor function score:emotion | baseline and 16, 28 weeks
  Hamilton Depression Scale to evaluate the degree of depression, Hamilton Anxiety Scale to evaluate the degree of anxiety
Non-motor function score:non-motor symptoms | baseline and 16, 28 weeks
  non-motor symptoms in PD patients is evaluated used Non-motor Symptoms Questionnaire
Non-motor function score:autonomic symptoms | baseline and 16, 28 weeks
  The scale for outcomes in PD for autonomic symptoms to assess autonomic dysfunction
Non-motor function score:the quality of life. | baseline and 16, 28 weeks
  The 39-item Parkinson's disease questionnaire to assess the quality of life.
Immunological index | baseline and 16, 28 weeks
  CD3(%)，CD4(%)，CD8(%)，Treg cells(%)
Imaging index | baseline and 16, 28 weeks
  Magnetic Resonance Imaging or positron emission tomography
Blood routine examination | baseline and 16, 28 weeks
  Blood routine examination includes the total number of red blood cells, hemoglobin, total number of white blood cells, white blood cells count, platelet count.
Biochemical routine examination | baseline and 16, 28 weeks
  Biochemical routine examination includes liver function, renal function, blood glucose, blood lipid
Safety index | 1,2,3,4,weeks and 16, 28 weeks
  Adverse Event and Serious Adverse Event

OTHER OUTCOMES:
PD therapy drugs | baseline and 16, 28 weeks
  Reduction rate of PD therapy drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Principal Investigator — Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Will decisde if the IPD based on patient consent

REFERENCES:
- [Result] Hallett PJ, Cooper O, Sadi D, Robertson H, Mendez I, Isacson O. Long-term health of dopaminergic neuron transplants in Parkinson's disease patients. Cell Rep. 2014 Jun 26;7(6):1755-61. doi: 10.1016/j.celrep.2014.05.027. Epub 2014 Jun 6. PMID 24910427
- [Result] Kefalopoulou Z, Politis M, Piccini P, Mencacci N, Bhatia K, Jahanshahi M, Widner H, Rehncrona S, Brundin P, Bjorklund A, Lindvall O, Limousin P, Quinn N, Foltynie T. Long-term clinical outcome of fetal cell transplantation for Parkinson disease: two case reports. JAMA Neurol. 2014 Jan;71(1):83-7. doi: 10.1001/jamaneurol.2013.4749. PMID 24217017